CLINICAL TRIAL: NCT05824403
Title: PAncreatic Disease Cohort of TOuLouse
Acronym: PACTOL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0530
Record Dates: First submitted 2023-03-27; First posted 2023-04-21 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Diseases
Keywords: Pancreatic cyst; Acute pancreatitis; chronic pancreatitis; Intra Pancreatic Mucinous Neoplasia; diagnosis
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Cyst; Pancreatitis; Pancreatitis, Chronic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective cohort dedicated to pancreatic diseases excluding cancer. The aim is to develop positive or differential diagnostic tools between benign potentially malignant or malignant pancreatic pathologies. During this study the investigators collect data and biological samples to support research project.

DETAILED DESCRIPTION:
This collection focuses on pathology of the pancreas requiring specific investigations or management for diagnosis or treatment. Pancreatic pathologies can be classified as malignant, potentially malignant or benign tumors. These can be solid or cystic. There is an inflammatory attack on the pancreas, generating acute pancreatitis in the acute period, if the inflammatory manifestations persist, chronic pancreatitis will develop. Some lesions may be at risk of malignancy during their evolution, it is therefore necessary to improve the performance of monitoring and diagnostic tools in order to adapt the management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory or cystic exocrine pancreatic pathology
* Patient able to read and understand the information leaflet
* Patients who have agreed to participate in the study and have signed the free and informed consent
* Patients affiliated to a social security system (including AME)

Exclusion Criteria:

* Patient with pancreatic cancer pathology
* Patients with active cancer, whatever the origin
* Pregnant or breastfeeding patients
* Patients under legal protection, guardianship or trusteeship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic tools | 3 years after the first inclusion
  To develop positive or differential diagnostic tools between benign potentially malignant or malignant pancreatic pathologies

SECONDARY OUTCOMES:
New targets | 3 years after the first inclusion
  To identify new screening targets
Improvement of management | 3 years after the first inclusion
  To improve the management of cystic lesions or Chronic pancreatitis on the decision of therapeutic management
Microbiota | 3 years after the first inclusion
  Study of the microbiota of pancreatic diseases
Clinical data access | 3 years after the first inclusion
  To make available to the scientific community quality material with associated clinical data also of quality

CONTACTS AND LOCATIONS:
Overall Officials: Barbara BOURNET, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Rangueil hospital, Toulouse, France

REFERENCES:
- [Derived] Bardol T, Dujon AM, Taly V, Dunyach-Remy C, Lavigne JP, Costa-Silva B, Kurma K, Eslami-S Z, Cayrefourcq L, Canivet C, Muscari F, Bournet B, Alix-Panabieres C. Early detection of pancreatic cancer by liquid biopsy "PANLIPSY": a french nation-wide study project. BMC Cancer. 2024 Jun 10;24(1):709. doi: 10.1186/s12885-024-12463-8. PMID 38853244